CLINICAL TRIAL: NCT02471612
Title: Comparative Analysis of APACHE II and P-POSSUM Scoring Systems in Predicting Postoperative Mortality in Patients Undergoing Emergency Laparotomy
Brief Title: Comparative Analysis of APACHE II and P-POSSUM
Status: Completed | Type: Observational
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Associate Specialist, Tata Main Hospital
Other Study IDs: 201-26104-132-108296
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2016-05

CONDITIONS: External Causes of Morbidity and Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare APACHE II and P-POSSUM scoring system in emergency laparotomy.

DETAILED DESCRIPTION:
To compare APACHE II and P-POSSUM scoring system in predicting postoperative mortality in patients undergoing emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years of age undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 will be included in the study.

Exclusion Criteria:

* Patients willingly seeking referral to a different hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 will be included in the study. All patients will be scored with APACHE II and P-POSSUM scoring systems on the day of surgery.The patients will be followed up till discharge, death or 30 days postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Dembla, DA, Principal Investigator — Tata Main Hospital, Jamshedpur, India
Locations (1):
- Tata Main Hospital, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nag DS, Dembla A, Mahanty PR, Kant S, Chatterjee A, Samaddar DP, Chugh P. Comparative analysis of APACHE-II and P-POSSUM scoring systems in predicting postoperative mortality in patients undergoing emergency laparotomy. World J Clin Cases. 2019 Aug 26;7(16):2227-2237. doi: 10.12998/wjcc.v7.i16.2227. PMID 31531317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, India who met the inclusion criteria were included in the study
Groups:
- All Patients Who Underwent Emergency Exploratory Laparotomy: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria were scored using the P-POSSUM Score APACHE-II
Period: Overall Study
Arm/Group | All Patients Who Underwent Emergency Exploratory Laparotomy
Started | 159
Completed | 157
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Emergency Laparotomy: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria were scored using the APACHE-2 Score & P-POSSUM Score
Arm/Group | Emergency Laparotomy
Number analyzed (Participants) | 157
Age, Customized [Number; unit: participants] — All patients above 18 years age were included in the study
  participants
    18- 20 years | 11
    21-40 years | 45
    41-60 years | 60
    61-80 years | 38
    > 80years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 99
Region of Enrollment [Number; unit: participants]
  India | 157

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Curve (ROC) as a Measure of the Accuracy of the APACHE II and P-POSSUM Scoring Systems to Predict Mortality
Description: Participants will be followed for the duration of hospital stay (expected average of 30 days) and mortality was noted.All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 were included in the study. All patients were scored with APACHE II and P-POSSUM scoring systems on the day of surgery. Area under the curve (AUC) is used to measure the "size" of the prediction composed by the graphic display between the 'sensitivity' and the '1-specificity' relationship. AUC can range from 0.5 to 1.0 and a result of 1.0 indicates a perfect discriminatory ability. An AUC value > 0.8 is considered good, a range between 0.60-0.80 is considered as moderate, and an AUC value < 0.60 is regarded as poor. For APACHE-II, a cut off score of >/=24 was determined; for P-POSSUM, a cut off score of >/= 63 was determined.
Time Frame: 30 days
Population: All patients undergoing emergency laparotomy at Tata Main Hospital form December 2013 to November 2014 were scored with APACHE II & P-POSSUM scoring systems on the day of surgery. The patients were followed up till at least 30 days after discharge or death (during admission or within 30 days after discharge).
Measure: Number (95% Confidence Interval); unit: probability of accurate prediction
Groups:
- AUC Using APACHE II: All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 were included in the study. All patients were scored with APACHE II on the day of surgery.
- AUC Using P-POSSUM: All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 were included in the study. All patients were scored with P-POSSUM on the day of surgery.
Arm/Group | AUC Using APACHE II | AUC Using P-POSSUM
Number analyzed (Participants) | 157 | 157
probability of accurate prediction | 0.965 [0.928 to 1.000] | 0.989 [0.974 to 1.000]
Statistical Analysis 1: Comparison: AUC Using APACHE II vs AUC Using P-POSSUM; Area under the curve (AUC) is used to measure the "size" of the prediction composed by the graphic display between the 'sensitivity' and the '1-specificity' relationship. AUC can range from 0.5 to 1.0 and a result of 1.0 indicates a perfect discriminatory ability. An AUC value > 0.8 is considered good, a range between 0.60-0.80 is considered as moderate, and an AUC value < 0.60 is regarded as poor; Test type: Superiority or Other; p = 0.665, McNemar — Comparing the sensitivity of APACHE-II and P-POSSUM

2. Secondary Outcome: Length of Stay (LOS)
Description: The mean duration of hospital stay or Length of Stay was recorded
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Length of Stay: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria were observed for their length of stay (LOS)
Arm/Group | Length of Stay
Number analyzed (Participants) | 157
Days
  Surviving Patients | 9.36 (8.04)
  Patients who Died | 14.91 (15.43)

3. Secondary Outcome: Need for Postoperative Ventilator Support
Description: Number of patients needing post-operative ventilatory support
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Surviving Patients: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and survived during the study period were observed if they needed ventilatory support postoperatively
- Patients Who Died: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and died during the study period were observed if they needed ventilatory support postoperatively
Arm/Group | Surviving Patients | Patients Who Died
Number analyzed (Participants) | 134 | 23
participants | 40 | 23

4. Secondary Outcome: Need for Post Operative Inotropic Support
Description: Number of patients needing post-operative inotropic support
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Surviving Patients: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and survived during the study period were monitored for the need for inotropic support during their stay..
- Patients Who Died: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and died during the study period were monitored for the need for inotropic support during their stay..
Arm/Group | Surviving Patients | Patients Who Died
Number analyzed (Participants) | 134 | 23
participants | 25 | 23

5. Secondary Outcome: Cardiac Morbidity (AMI or Arrhythmias Needing Treatment)
Description: Number of patients noted to have Cardiac morbidity: Acute myocardial infarction (AMI) or arrhythmias needing treatment
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Patients Who Survived: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and survived during the study period were monitored for Cardiac morbidity (Acute Myocardial Infarction (AMI) or arrhythmias needing treatment)
- Patients Who Died: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and died during the study period were monitored for Cardiac morbidity (Acute Myocardial Infarction (AMI) or arrhythmias needing treatment)
Arm/Group | Patients Who Survived | Patients Who Died
Number analyzed (Participants) | 134 | 23
participants | 1 | 7

6. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI)
Description: Acute Kidney Injury (AKI) was diagnosed based on the Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group (2012) guidelines
  1. Increase in Serum Creatinine (S. Cr) by ≥0.3 mg/dl (≥ 26.5 μmol/l) within 48 hours; OR
  2. Increase in S. Cr to ≥1.5 times baseline, which is known or presumed to have occurred within prior 7 days; OR
  3. Urine volume <0.5 ml/kg/h for 6 hours
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Patients Who Survived: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and survived during the study period were monitored for the Acute Kidney Injury
- Patients Who Died: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and died during the study period were monitored for the Acute Kidney Injury
Arm/Group | Patients Who Survived | Patients Who Died
Number analyzed (Participants) | 134 | 23
participants | 14 | 18

7. Secondary Outcome: Patients Needing Re-exploration
Description: Number of patients needing return to the operation theater for surgery for the same pathology or any other complication arising out of the initial surgery
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Patients Who Survived: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and survived during the study period were observed if they needed re-exploration during the post-operative period.
- Patients Who Died: All patients who underwent emergency exploratory laparotomy from December 2013 to November 2014 at the Tata Main Hospital, Jamshedpur, and met the inclusion criteria and died during the study period were observed if they needed re-exploration during the post-operative period.
Arm/Group | Patients Who Survived | Patients Who Died
Number analyzed (Participants) | 134 | 23
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: The patients were followed up for the duration of admission and till at least 30 days after discharge or death (whichever was earlier).
Groups:
- APACHE-2 Scoring: All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 were included in the study. All patients were scored with APACHE II on the day of surgery.
- P-POSSUM: All patients undergoing emergency laparotomy at Tata Main Hospital form 01st December 2013 to 30th November 2014 were included in the study. All patients were scored with P-POSSUM on the day of surgery
Arm/Group | APACHE-2 Scoring | P-POSSUM
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157

LIMITATIONS AND CAVEATS:
Observational study. So no specific adverse effect because of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes